CLINICAL TRIAL: NCT07367464
Title: Radiographic And Histomorphometric Assessment Of Guided Bone Regeneration Using Xenograft Mixed With Allogenic Bone Graft Versus Xenograft Mixed With Autogenous Bone Graft For Augmentation Of Deficient Maxillary Alveolar Ridges A Randomized Clinical Trial
Brief Title: Assessment Of Guided Bone Regeneration Using Xenograft Mixed With Allogenic Bone Graft Versus Xenograft Mixed With Autogenous Graft For Augmentation Of Maxillary Alveolar Ridges
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdulnaser Abousetta, Master Degree student, Implantology department, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-5-24
Record Dates: First submitted 2026-01-14; First posted 2026-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Guided Bone Regeneration
Keywords: Guided Bone Regeneration; DFDBA; Autogenous Bone Graft; Xenograft; Xenograft Mixed With Autogenous Bone Graft; Xenograft Mixed With Allogenic Bone Graft; Deficient Maxillary Alveolar Ridges
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of the participants and the operator is not applicable, however outcome assessors and bio-statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogenic bone graft mixed with Xenograft in ratio 1:1 (Experimental): A full thickness flap will be elevated with two releasing incisions extending at least just distal to each tooth adjacent to the defect site.The flap will be reflected adequately to expose the defect. The cortical bone will be perforated with a small round bur to perform decortication of the buccal aspect of the ridge. recipient site will be debrided from any soft tissue or periosteum remnants.The grafts will be placed on the buccal aspect of the alveolar ridge, layer by layer, gently pressed to the recipient site then it will be covered by a collagen pericardium membranes. The membrane will be stretched tightly over the graft and titanium tacks will be placed at the labial side to fix the membrane in place. The incisions will be carefully closed with horizontal mattress sutures as well as single interrupted and continuous with resorbable sutures.
  Interventions: Biological: Allogenic bone graft mixed with Xenograft in ratio 1:1
- Autologous bone graft mixed with Xenograft in ratio 1:1 (Active Comparator): A full thickness flap will be elevated with two releasing incisions extending at least just distal to each tooth adjacent to the defect site.The flap will be reflected adequately to expose the defect. The cortical bone will be perforated with a small round bur to perform decortication of the buccal aspect of the ridge. recipient site will be debrided from any soft tissue or periosteum remnants.The grafts will be placed on the buccal aspect of the alveolar ridge, layer by layer, gently pressed to the recipient site then it will be covered by a collagen pericardium membranes. The membrane will be stretched tightly over the graft and titanium tacks will be placed at the labial side to fix the membrane in place. The incisions will be carefully closed with horizontal mattress sutures as well as single interrupted and continuous with resorbable sutures.
  Interventions: Biological: Autologous bone graft mixed with Xenograft in ratio 1:1

INTERVENTIONS:
Biological: Allogenic bone graft mixed with Xenograft in ratio 1:1 — Xenogenic graft is then to be mixed in equal 1:1 volume of particles size 0.25-1 mm with the Allogenic bone graft chips to create 1:1 composite graft.
  Arms: Allogenic bone graft mixed with Xenograft in ratio 1:1
Biological: Autologous bone graft mixed with Xenograft in ratio 1:1 — Autogenous bone particulate will be harvested either from the mandibular symphysis or ramus. Mandibular symphysis as a donor site: A beveled partial to full thickness muco-periosteal incision 5 to 10 mm below the muco-gingival junction will be performed at the symphyseal region to expose the donor site. The incision extended just distal to the mandibular canines to allow for adequate access and easier adaptation of the flap.Mandibular ramus as a donor site: A submarginal incision will be placed within the keratinized mucosa opposite to the lower first molar and extending 1 cm along the ramus of the mandible.
  Arms: Autologous bone graft mixed with Xenograft in ratio 1:1

SUMMARY:
This study aims to evaluate the effect of Allogenic bone graft mixed with Xenograft in ratio 1:1, on the radiographic and histomorphometric assessment versus Autologous bone graft mixed with Xenograft in ratio 1:1 in maxillary deficient ridges، In guided bone regeneration of deficient edentulous maxillary ridges, will the application of Xenograft mixed with Allograft (1:1) be as effective as Xenograft mixed with Autogenous graft (1:1) in terms of dimensional ridge changes and Quality of newly formed bone?

Evaluation of the patient's general condition of the oral cavity, to make sure it complies with the criteria required to be enrolled in the study in terms of oral hygiene and pathological conditions.

A full thickness flap will be elevated with two releasing incisions, decortication of the buccal aspect of the ridge, placing of grafting material which will be covered by collagen pericardium membranes, tacks placement at the labial side to fix the membrane in place, horizontal mattress sutures as well as single interrupted and continuous with resorbable sutures for closure.

Intervention group: will be filled with mixture of Xenogenic graft and the Allogenic bone graft chips.

Control group: will be filled with mixture of Xenogenic graft and Autogenous bone particulate harvested either from the mandibular symphysis or ramus.

For both groups, All the subjects will be taking CBCT at pre surgical and 6 months post surgical. outcomes : Bucco-Palatal/Lingual horizontal bone gain, Alveolar ridge height,Percentage of new vital bone formation and Percentage of residual bone graft 6 months post-surgical.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of Allogenic bone graft mixed with Xenograft in ratio 1:1, on the radiographic and histomorphometric assessment versus Autologous bone graft mixed with Xenograft in ratio 1:1 in maxillary deficient ridges. Null hypothesis: no significant difference in ridge dimensional changes is expected to occur on comparing Xenograft mixed with Allograft versus Xenografts mixed with autogenous bone grafts in guided bone regeneration.

The study will be conducted at the post-graduate clinic of the periodontology and Oral Implantology Departments, Faculty of Dentistry, Cairo University, Egypt. Patients will be selected from the outpatient clinic of the Department of Oral Implantology, Cairo University.

1. Clinical examination & informed consent: Evaluation of the patient's general condition of the oral cavity, to make sure it complies with the criteria required to be enrolled in the study in terms of oral hygiene and pathological conditions.
2. Radiographic examination: Preoperative cone beam computed tomography (CBCT) will be done to exclude any pathosis and measure the bone width of the deficient area. Bone width will be measured from the reformatted cross-sectional image of the CBCT 2.0 mm below the tip of the crest at every single deficient site taking a specific anatomical landmark in the opposing teeth as a reference point for the measurements taking into consideration that the patients are biting in maximum intercuspation. The average of these measurements will be calculated to be a representative value of the preoperative width for each case from the preoperative CBCT. Immediate and 6 months postoperative CBCT will be done with the patients biting in maximum intercuspation and the same measurements will be taken from the same reference areas that were previously selected from the preoperative scan. Alveolar height will be measured from crest of the ridge to the nasal floor or sinus floor.
3. Surgical procedures: Local anesthesia will be administered by infiltration or nerve block to achieve the necessary anesthesia and guided bone regeneration will be done according to the allocation concealment.All procedures will be performed by the same surgeon.As a prophylactic measure all patients will receive 2 g of V-penicillin amoxicillin/clavulanate 2 g for 10 days starting 1 hour pre-operatively or Clindamycin 300 mg for 10 days in event of penicillin allergy.

   A full thickness flap will be elevated with two releasing incisions extending at least just distal to each tooth adjacent to the defect site. vertical incisions at the canine eminence will be avoided and instead extended distal to the canine to avoid future dehiscence at this site. The flap will be reflected adequately to expose the defect. The cortical bone will be perforated with a small round bur to perform decortication of the buccal aspect of the ridge.

   Control group (Xenograft + Autogenous bone) Autogenous bone particulate will be harvested either from the mandibular symphysis or ramus.

   A. Mandibular symphysis as a donor site:

   A beveled partial to full thickness muco-periosteal incision 5 to 10 mm below the muco-gingival junction will be performed at the symphyseal region to expose the donor site. The incision extended just distal to the mandibular canines to allow for adequate access and easier adaptation of the flap.

   B. Mandibular ramus as a donor site:

   A submarginal incision will be placed within the keratinized mucosa opposite to the lower first molar and extending 1 cm along the ramus of the mandible.

   For both donor sites, autogenous bone will be harvested by an Auto-chip maker (ACM) bur and the harvested Autogenous bone chips is then to be mixed in equal ratio 1:1 volume with Xenograft of particle size 0.25-1 mm and will be added to the harvested autogenous bone to create 1:1 composite graft.

   Intervention group (Xenograft + Allograft) Xenogenic graft is then to be mixed in equal 1:1 volume of particles size 0.25-1 mm with the Allogenic bone graft chips 0.25-1mm to create 1:1 composite graft.

   The recipient site will be debrided from any soft tissue or periosteum remnants. The grafts will be placed on the buccal aspect of the alveolar ridge, layer by layer, gently pressed to the recipient site. All grafts will be covered by a collagen pericardium bio-resorbable membranes. The membrane will be stretched tightly over the graft and titanium tacks will be placed at the labial side to fix the membrane in place. Additional particulate will be packed under the membrane laterally to over fill the site. With bone tack pin fixation at both lingual and buccal sides. The particulate composite graft will be packed onto the defect and overfilling will be done to compensate for future resorption.The incisions will be carefully closed with horizontal mattress sutures as well as single interrupted and continuous with resorbable sutures.

   Follow-up protocol will be done every other day for the first week, weekly for the first month, and then monthly for 3 months. Postoperative CBCT scans will be done for all patients at 6 months interval, to assess the amount of horizontal bone gain which is the primary outcome.
4. Second stage surgery:

   After 6 months, re-entry will be done utilizing a full thickness mucoperiosteal flap, and a core biopsy will be taken using a 2 mm trephine bur from the pre-planned implant positions in the direction of the implant osteotomy for histomorphometric analysis of the augmented bone to measure the bone area percent which is the secondary outcome. Dental implants with diameters ranging 3.7 to 4.2 mm will be inserted in the augmented ridge in a 2-stage procedure according to the manufacturer's protocol. Cover screws will be placed, and the flaps will be adapted with resorbable 4-0 sutures.
5. Histomorphometric and statistical analysis:

   The core biopsies will be sectioned and stained with H&E stain for examination under a light microscope with a ×50 magnification. Bone volume will be measured for each specimen and the mean volume for native bone and newly formed bone will be calculated for statistics.Quantitative histomorphometric analysis will be performed by OLYMPUS Stream software. Data management and statistics will be done by using the Statistical Package for Social Sciences version 22.
6. Postoperative instructions and follow up:

   Antibiotics (Amoxicillin 1g twice daily for 5 days) to prevent postoperative infection.Anti-inflammatory drugs (NSAIDS; Ibuprofen 600mg three times daily for 5 days) to avoid edema, pain or swelling.Antiseptic mouth rinse (0.12% Chlorhexidine oral rinse will be prescribed for 60 seconds two times a day for 14 days.
7. Patient self-care instructions:

Patients will be instructed to apply an ice bag to the treated area for the first 24 hours and avoid any brushing and trauma to the surgical site for one week.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-60 years.
* Totally or partially edentulous maxillary ridges.
* Patients with insufficient bone for an implant placement.
* Residual alveolar width ranging from 2 to 4 mm.
* Minimum of 10 mm vertical dimension to nasal floor or sinus floor.
* Patients with healthy systemic condition (Medically free).
* Adequate inter-arch space for placement of the implant prosthetic part.

Exclusion Criteria:

* Pathological lesions in the defect site.
* Systemic diseases that would interfere with bone metabolism. Uncontrolled diabetic patients.
* Ongoing treatment or a history of recent chemotherapy or radiotherapy.
* Patient with medical condition that contraindicates surgical procedures.
* Patients on medication that may interfere with healing (Corticosteroids, Bisphosphonate, Chemo/radio therapy).
* Patients with vertical bone deficiency.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as alcoholism or para-functional habits.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Bucco-Palatal/Lingual horizontal bone gain | 6 months postoperatively
  Bone width will be measured from the reformatted cross-sectional image of the CBCT 2 mm below the tip of the crest at every single deficient site taking a specific anatomical landmark in the opposing teeth as a reference point for the measurements taking into consideration that the patients are biting in maximum intercuspation. The average of these measurements will be calculated to be a representative value of the preoperative width for each case from the preoperative CBCT. Immediate and 6 months postoperative CBCT will be done while the patients are also biting in maximum intercuspation and the same measurements will be taken from the same reference areas previously selected from the preoperative scan.

SECONDARY OUTCOMES:
Alveolar ridge height: | 6 months postoperatively
  It will be measured from the crest of the ridge to the nasal floor or sinus floor.
Percentage of new vital bone formation | 6 months postoperatively
  core biopsies will be preserved in a 10% formalin solution. Following that, they will undergo four weeks of EDTA decalcification. The specimens will be treated and embedded in paraffin after decalcification to generate tissue blocks. The paraffin blocks will be split into longitudinal sections of 5m thickness. For histological examination and histomorphometric analysis, these slices will be stained with hematoxylin and eosin (H&E) or Masson's trichromatic (MT) stains. A digital light microscope will be used to photograph the stained sections.
  Histomorphometric analysis will be undertaken to determine the percentage of the total analysed histological area occupied by bone, graft particles, and soft tissue stroma using (Leica QWin 500 image analysis software, Leica Microsystems, Switzerland).
Percentage of residual bone graft | 6 months postoperatively
  core biopsies will be preserved in a 10% formalin solution. Following that, they will undergo four weeks of EDTA decalcification. The specimens will be treated and embedded in paraffin after decalcification to generate tissue blocks. The paraffin blocks will be split into longitudinal sections of 5m thickness. For histological examination and histomorphometric analysis, these slices will be stained with hematoxylin and eosin (H&E) or Masson's trichromatic (MT) stains. A digital light microscope will be used to photograph the stained sections. Histomorphometric analysis will be undertaken to determine the percentage of the total analysed histological area occupied by bone, graft particles, and soft tissue stroma using (Leica QWin 500 image analysis software, Leica Microsystems, Switzerland).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Abousetta, Bachelor, Principal Investigator — Cairo University; Mohamed M. Shaker, Professor, Study Chair — Cairo University; Weam A. El-Battawy, Ass. Prof., Study Director — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt